CLINICAL TRIAL: NCT03725527
Title: Respiratory Effects of Rectus Sheath Block in Patients Undergoing Major Upper Abdominal Surgery.
Brief Title: Effect of Rectus Sheath Block on Diaphragmatic Function After Elective Upper Abdominal Surgery
Acronym: Rectus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noha Yahia Mohammd El-hagagy, Lecturer of anesthesia and intensive care, faculty of medicine, Assiut university., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17100594
Record Dates: First submitted 2018-09-29; First posted 2018-10-31 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectus sheath block (Active Comparator): Patients will receive ultrasound-guided rectus sheath block' performed after induction of general anesthesia and before surgery.
  Interventions: Procedure: Rectus Sheath Block
- control (No Intervention): Patients will receive general anesthesia .

INTERVENTIONS:
Procedure: Rectus Sheath Block — Sonar guided RSB will be performed using a 16-G, 8-cm TuohyUpon reaching this potential space, after careful aspiration.
  Other Names: RSB
  Arms: Rectus sheath block

SUMMARY:
This study will be undertaken to investigate the respiratory and analgesic effects of ultrasound guided rectus sheath block analgesia after elective abdominal surgery with midline incision.

DETAILED DESCRIPTION:
A major proportion of pain experienced by patients undergoing abdominal surgeries is due to somatic pain signals derived from the abdominal wall. The central portion of anterior abdominal wall components (skin, muscles and parietal peritoneum) is innervated by sensory neurons branching from the anterior rami of spinal nerves T7 to T1. These neurons lie between the rectus abdominis muscle and posterior rectus sheath, and pierce the rectus muscle close to the midline. The tendinous intersections of the rectus muscle do not fuse with the posterior rectus sheath, thereby allowing the injectate to spread cephalo-caudally within this potential space. Rectus sheath (RS) block has been described for any midline abdominal incisions (epigastric and umbilical hernia repairs). As visceral pain becomes attenuated by the 2nd postoperative day, rectus sheath block can also be administered for midline laparotomy.

However, the effects of rectus sheath block analgesia on the respiratory function after abdominal surgery with midline incisions are still under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-50 years.
* Sex: both males and females.
* BMI< 30kg/m2.
* ASA physical status: 1, II and III.
* Elective abdominal surgery with midline incisions.

Exclusion Criteria:

* Patient refusal.
* Infection at injection site
* Coagulation disorders.
* Allergy to study medications.
* Pregnancy.
* Respiratory tract infection within the last 2 weeks.
* Urgent abdominal surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic inspiratory amplitude during quiet/deep breathing (DIA)/cm | 24 hours Postoperative
  The ultrasonic measurements of diaphragmatic motion will be attained at the posterior surface of the diaphragm. From the tracings on M-mode, the distance between echogenic lines (DIA) in centimeters and diaphragmatic inspiratory/expiratory velocity in centimeters/second during quiet, deep, and sniff breathing will be measured on the frozen images.

SECONDARY OUTCOMES:
Verbal Rating Scale | 24 hours Postoperatively
  Verbal rating pain scale (VRS) (Ranging from 0 to 4), where 0=no pain, 1=mild pain, 2=moderate pain, 3=severe pain and lastly 4 =excruciating pain) will be recorded at rest and upon patient coughing; on admission to PACU (baseline), and 2, 4, 6, 12, and 24h postoperatively.
Forced Vital Capacity/L | 24 hours Postoperatively
  Measurements of Forced vital capacity (FVC) will be measured by the use of hand-held spirometer (One-flow®, Clement Clarke, U.K). At each assessment, the largest values of FVC will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Y Mohamed, MD, Principal Investigator — Lecturer in anesthesia and intensive care department, faculty of medicine, Assiut university, Egypt.
Locations (1):
- Assiut university main hospital, ICUs, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No